CLINICAL TRIAL: NCT04814563
Title: Evaluation of the Contribution of Comparative Genomic Hybridization Compared to Karyotype for the Detection of Genetic Abnormalities According to Ultrasound Call Signs in Prenatal Screening: the Cohort of the Nancy Multidisciplinary Center for Prenatal Diagnosis From 2012 to 2018
Brief Title: Evaluation of the Relevance of Comparative Genomic Hybridization in Prenatal Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, PERDRIOLLE-GALET Estelle, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI288
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Comparative Genomic Hybridization
Keywords: Prenatal diagnosis; Ultrasound sign

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pre-natal diagnosis is developing nowadays thanks to the improvement of ultrasound performances but also of genetic analysis techniques.

The karyotype was previously the reference technique for genetic analysis. The development of comparative genomic hybridization, consisting of comparative genomic hybridization on DNA sequences and allowing the diagnosis of unbalanced chromosomal rearrangements, has made it possible to increase the resolution threshold for the detection of genetic anomalies. This technique can be performed both pre and post natal. In pre-natal, the indications for this genetic study are based on ultrasound signs and are regularly updated in the international literature. Due to the complete analysis of the genome and the increase of the resolution threshold, genetic anomalies not related to the detected ultrasound pathology may be discovered and may pose ethical problems from a genetic counseling point of view.

To date, the diagnostic performance of comparative genomic hybridization as a complement to karyotype is being confirmed and needs to be clarified in order to limit the risk of incidental discovery of genetic anomalies whose significance remains unknown.

Through the study that the investigator would like to carry out, the investigator seek to evaluate the diagnostic contribution of this comparative genomic hybridization technique compared to the data provided by the karyotype according to the various ultrasound call signs on the Nancy cohort of files presented to the multidisciplinary pre-natal diagnosis committee, since the launch of the comparative genomic hybridization in Nancy in 2012 until 2018.

ELIGIBILITY:
Inclusion Criteria:

* CGH-array performed for ultrasound findings at the genetic laboratory of the Nancy University Hospital from 01/10/2012 to 31/12/2018
* Results of the CGH-array presented to the multidisciplinary pre-natal diagnosis committee of Nancy

Exclusion Criteria:

* patients who objected to the use of their data for research purposes when signing the informed consent form given during the genetic consultation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent amniocentesis or chorionic villus puncture during their pregnancy due to ultrasound call sign with CGH-array performed at the Nancy University Hospital genetics laboratory
Sampling Method: Non-Probability Sample
Enrollment: 830 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
CGH-array abnormality | baseline
  An anomaly will be detected at CGH-array if its size is greater than or equal to 500 Kb. Size of these anomalies will be considered in a binary manner: < 10 Mb (i.e. not visible on karyotype) and ≥ 10 Mb (i.e. visible on karyotype)

SECONDARY OUTCOMES:
Type of ultrasound call sign | baseline
  The ultrasound signs will be defined by the ultrasound technician thanks to the recommended classification
Genotype-phenotype concordance | baseline
  The genotype-phenotype concordance is defined by the cytogeneticist who delivers the results, according to the current scientific knowledge described in the literature
Particular gravity | baseline
  The particular gravity (Yes/No) of the ultrasound sign is defined after consultation between the various health professionals gathered at the multidisciplinary pre-natal diagnosis committee (gynaecologist, paediatrician, geneticist, radiologist, histopathologists, surgeons, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Estelle PERDRIOLLE-GALET, Doctor, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Nancy University Hospital, Nancy, France

REFERENCES:
- [Background] Rudolf G, Lovrecic L, Tul N, Teran N, Peterlin B. The frequency of CNVs in a cohort population of consecutive fetuses with congenital anomalies after the termination of pregnancy. Mol Genet Genomic Med. 2019 Jun;7(6):e658. doi: 10.1002/mgg3.658. Epub 2019 Apr 19. PMID 31004418
- [Background] Stosic M, Levy B, Wapner R. The Use of Chromosomal Microarray Analysis in Prenatal Diagnosis. Obstet Gynecol Clin North Am. 2018 Mar;45(1):55-68. doi: 10.1016/j.ogc.2017.10.002. Epub 2017 Dec 9. PMID 29428286
- [Background] Lo JO, Shaffer BL, Feist CD, Caughey AB. Chromosomal microarray analysis and prenatal diagnosis. Obstet Gynecol Surv. 2014 Oct;69(10):613-21. doi: 10.1097/OGX.0000000000000119. PMID 25336071
- [Background] Lee CN, Lin SY, Lin CH, Shih JC, Lin TH, Su YN. Clinical utility of array comparative genomic hybridisation for prenatal diagnosis: a cohort study of 3171 pregnancies. BJOG. 2012 Apr;119(5):614-25. doi: 10.1111/j.1471-0528.2012.03279.x. Epub 2012 Feb 7. PMID 22313859
- [Background] Wou K, Levy B, Wapner RJ. Chromosomal Microarrays for the Prenatal Detection of Microdeletions and Microduplications. Clin Lab Med. 2016 Jun;36(2):261-76. doi: 10.1016/j.cll.2016.01.017. Epub 2016 Mar 28. PMID 27235911
- [Background] Levy B, Wapner R. Prenatal diagnosis by chromosomal microarray analysis. Fertil Steril. 2018 Feb;109(2):201-212. doi: 10.1016/j.fertnstert.2018.01.005. PMID 29447663
- [Background] Wapner RJ, Martin CL, Levy B, Ballif BC, Eng CM, Zachary JM, Savage M, Platt LD, Saltzman D, Grobman WA, Klugman S, Scholl T, Simpson JL, McCall K, Aggarwal VS, Bunke B, Nahum O, Patel A, Lamb AN, Thom EA, Beaudet AL, Ledbetter DH, Shaffer LG, Jackson L. Chromosomal microarray versus karyotyping for prenatal diagnosis. N Engl J Med. 2012 Dec 6;367(23):2175-84. doi: 10.1056/NEJMoa1203382. PMID 23215555